CLINICAL TRIAL: NCT01003366
Title: Effect of the Bevel Direction of Puncture Needle on Success Rate and Complications During Central Venous Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Hyon Bahk, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: JHBahk_CVC bevel
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Central Venous Catheterization
Keywords: safety during central venous catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bevel down (Experimental): approaching the IJV with the needle bevel facing down
  Interventions: Device: bevel direction during central venous catheterization
- bevel up (Active Comparator): approaching the IJV with the needle bevel facing up
  Interventions: Device: bevel direction during central venous catheterization

INTERVENTIONS:
Device: bevel direction during central venous catheterization — approaching the IJV with the needle bevel facing down
  Arms: bevel down
Device: bevel direction during central venous catheterization — approaching the IJV with the needle bevel facing up
  Arms: bevel up

SUMMARY:
To test the hypothesis that approaching the internal jugular vein with the needle bevel down would produce less injury to the vessel wall compared to the bevel up approach during central venous catheterization.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery that requires the placement of a central venous catheter at the internal jugular vein

Exclusion Criteria:

* anatomical anomaly in the neck region
* recent history of central venous catheterization

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
posterior wall puncture of internal jugular vein | immediately after catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea